CLINICAL TRIAL: NCT01457820
Title: Allopurinol as a Possible New Therapy for Acute Coronary Syndromes:The Next Steps
Brief Title: Allopurinol in Acute Coronary Syndrome
Acronym: ALLACS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment: stopped early
Sponsor: Stephen McSwiggan (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, Stephen McSwiggan, Senior Clinical Trials Manager, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010CV30
Record Dates: First submitted 2011-10-17; First posted 2011-10-24 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Stable Angina
Keywords: Allopurinol; Angina; Acute coronary syndrome
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Acute Coronary Syndrome | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Allopurinol High dose (Experimental)
  Interventions: Drug: Allopurinol
- Allopurinol Low dose (Experimental)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Stat dose Allopurinol 800mg, then 400mg BD for 5 days
  Arms: Allopurinol High dose
Drug: Allopurinol — Stat dose Allopurinol 400mg, then 300mg BD for 5 days
  Arms: Allopurinol Low dose
Drug: Placebo — Matched placebo, stat dose, then 5 days of matched placebo BD.
  Arms: Placebo

SUMMARY:
Allopurinol is a drug commonly used to treat gout. However recent studies have shown it has the potential to help improve oxygen supply to heart muscle. In this study the Investigators aim to find out if allopurinol slows down the onset of angina symptoms, as seen by a doctor on a tracing of the heart (ECG- electrocardiogram), for patients who have been diagnosed with heart disease, when exercising on a treadmill. The Investigators are also are trying to figure out the best dose of allopurinol to use and to see how quickly it begins working. To do this the investigators will recruit patients with angina, exercise them on a treadmill after giving different doses of allopurinol and see if there is an improvement in their time to bring on angina symptoms and signs. Patients recruited to this trial will receive three different treatment regimes over a six week period. Each treatment regime will last for one week with a one week rest period between each regime. This will involve up to eleven visits to Ninewells Medical School, Dundee for testing.

ELIGIBILITY:
Inclusion Criteria:

* angiographically documented coronary artery disease,
* a positive exercise tolerance test (ETT)
* a history of symptoms of chronic, stable, effort-induced angina for ≥ 2 months.
* All concomitant antianginal medication will be allowed and continued unchanged during the study.

Exclusion Criteria:

* the inability to do an ETT due to back or leg problems,
* myocardial infarction or acute coronary syndrome ≤ 2 months,
* coronary revascularization (percutaneous or CABG) ≤ 6 months,
* Left Ventricular Ejection Fraction <45%,
* estimated GFR <60 ml/min or creatinine >180 mmol/ml,
* significant valvular pathology,
* already had gout or on allopurinol,
* atrial arrhythmias or ECG abnormalities interfering with ST-segment interpretation,
* previous ventricular arrhythmias on ETT,
* severe hepatic disease
* or on azathioprine, 6 mercaptopurine or warfarin.
* Patients who have participated in any other clinical trial within the previous 30 days will be excluded.
* Patients who are unable to give informed consent will also be excluded from this trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in time to exercise induced ST depression | 4 hours, 1 day and 5 days post study drug testing compared to Baseline 1 hour pre study drug
  A continuous ECG tracing will be recorded. Time to >1mm change in ST measurements will be noted. Exercise Tolerance testing (ETT) 1 hour before study drug administration is baseline measurement. Comparisons will be made 4 hours, 1 day and 5 days after baseline ETT.

SECONDARY OUTCOMES:
change in total exercise time on Exercise Tolerance Testing (ETT) | 4 hours, 1 day and 5 days post study drug testing compared to Baseline 1 hour pre study drug
  A continuous ECG tracing will be recorded. Time to total exercise time, ie when patient can walk no further will be noted. Exercise Tolerance Testing (ETT) 1 hour before study drug administration is baseline measurement. Comparisons will be made 4 hours, 1 day and 5 days after baseline ETT.
Change in time to subjects reported symptoms of chest pain during exercise testing. | hours, 1 day and 5 days post study drug testing compared to Baseline 1 hour pre study drug
  A continuous ECG tracing will be recorded. Time to reported chest pain will be noted. Exercise Tolerance testing (ETT) 1 hour before study drug administration is baseline measurement. Comparisons will be made 4 hours, 1 day and 5 days after baseline ETT.
changes in blood markers, specifically Brain Naturetic Peptide (BNP), high sensitivity Troponin T and high sensitivity C Reactive Protein (hsCRP), during exercise testing | Pre and post 4 hour ETT compared to baseline
  Baseline is pre 1st study drug dose exercise tolerance test (ETT). Comparisons will be made before and after 4 hour post drug ETT
angina pain and Glyceryl TriNitrate (GTN) usage | Weekly
  subjects will use angina log to record symptoms of angina and GTN usage between hospital visits

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, BSc, MD, FRCP, FRSE, FMedSci, Principal Investigator — University of Dundee
Locations (1):
- NHS Tayside, Dundee, Angus, United Kingdom